CLINICAL TRIAL: NCT00269243
Title: The Ischemia Management With Accupril Post Bypass Graft Via Inhibition of the coNverting Enzyme (IMAGINE) Trial
Brief Title: Management With Accupril Post Bypass Graft
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: IMAGINE ID: 906-437
Record Dates: First submitted 2005-12-20; First posted 2005-12-23 (Estimated); Last update posted 2006-02-08 (Estimated); Status verified 2005-12

CONDITIONS: CABG
MeSH Terms: interventions — Quinapril

INTERVENTIONS:
Drug: Quinapril

SUMMARY:
Angiotensin converting enzyme (ACE) inhibitors have been shown to improve survival and to reduce the risk of cardiovascular events in some groups of patients following myocardial infarction. This study is designed to test whether early initiation (≤7 days) of an ACE inhibitor post-coronary artery bypass graft (CABG), would reduce cardiovascular events. The trial was a double-blind, placebo controlled study of 2,553 patients randomly assigned to quinapril, target dose 40 mg daily or placebo, followed up to 43 months.

DETAILED DESCRIPTION:
The IMAGINE study is a double-blind, placebo controlled, parallel group, randomized, multi-centre international study conducted in patients who have undergone CABG. The research protocol was approved by the ethics committee of all participating institutions, and all patients gave written informed consent. The data were collected and analysed by an independent clinical research organization.

Patients were screened for eligibility and randomized in hospital within seven days post-CABG, except for France where randomization could occur within ten days post-CABG. Starting November 6, 2001, given the increasing evidence of benefit of ACE inhibitors in patients with diabetes and renal disease,14 all patients requiring insulin or with type II diabetes and micro-albuminuria were no longer eligible for the study. Those already in the trial were treated according to the clinical judgement of the treating physician.

Of patients screened in 57 sites in Canada, the Netherlands, Belgium or France, 2 553 patients (approximately 5 percent of patients screened) were randomized post-operatively to quinapril either 10 or 20 mg, or to placebo. Randomization was done centrally, was un-stratified, block-based, and computer generated. If tolerated, patients were up-titrated to 40 mg of quinapril or its placebo equivalent within hospital, or if not tolerated, later post-hospital discharge. Patients were followed for twenty-four months at which time they were invited to continue until 43 months of follow-up, or withdrawn if they did not wish to extend their participation in the trial.

The original primary endpoint consisted of time to first occurrence of any of the composite of cardiovascular death or resuscitated cardiac arrest, nonfatal myocardial infarction, coronary revascularization, unstable angina requiring hospitalization and documented angina not requiring hospitalization. On January 14, 2003, the Steering Committee concluded that the required number of endpoints would likely not be reached without modification of the primary endpoint. Stroke and congestive heart failure requiring hospitalization were thus added to the primary endpoint and sample-size was increased to 2 500 patients.

The secondary endpoints included, 1) time to first occurrence of the following composite of cardiovascular death or resuscitated cardiac arrest, nonfatal myocardial infarction, coronary revascularization or stroke; 2) incidence of any of the above mentioned secondary endpoints; 3) time to first occurrence of the composite primary endpoint with the addition of the following: transient ischemic attack, and any cardiovascular event requiring hospitalization; 4) incidence of any secondary endpoints included in #3; and 5) time to occurrence of death from any cause. All endpoints were adjudicated in a blinded fashion by an endpoint committee, based on pre-defined definitions for each endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Post-CABG less than or equal to 7 days (10 days in France)
* Stable post-operation (as per investigator judgement)
* Still in hospital
* 18 years of age or older
* LVEF ≥40 percent determined within six months before surgery

Exclusion Criteria:

* Intolerance/contraindication to ACE-inhibitor or history of angioedema
* Insulin-dependent diabetes, or type II diabetes with microalbuminuria
* Clinical need for an ACE inhibitor or an angiotensin receptor blocker (investigators' judgement)
* Current need for post-CABG urgent intervention
* Valve replacement, not repair, during index CABG
* Significant valve stenosis or cardiomyopathy
* Serum potassium concentration of 5.6 mmol per liter or more
* Primary hyperaldosteronism
* Serum creatinine greater than 2.26 mg per decilitre (suspected renal artery stenosis, single kidney or renal transplant
* Serious concomitant disease, such as cancer, AIDS, sepsis
* SBP >160 mm Hg or DBP <90 mm Hg despite treatment
* SBP <100 mm Hg
* Significant peri-operative myocardial infarction
* Pregnancy, breastfeeding, inadequate contraception
* Investigational drug use <30 days
* Drug, alcohol abuse, inability to adhere to protocol.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 1999-11; Study Completion 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Lucien Rouleau, M.D, Principal Investigator — Montreal Heart Institute